CLINICAL TRIAL: NCT06300242
Title: Financial Incentives for Influenza Vaccination
Brief Title: Incentives for Influenza Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: J-PAL North America (Unknown)
Responsible Party: Principal Investigator, Mireille Jacobson, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UP-23-00859
Record Dates: First submitted 2024-02-28; First posted 2024-03-08 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Influenza Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Message Only (Experimental): Patients sent an email or SMS reminding them to get vaccinated against the flu.
  Interventions: Behavioral: Reminders
- Message + Financial Incentive (Experimental): Patients sent an email or SMS reminding them to get vaccinated against the flu and offering them a $50 financial incentive if they are vaccinated within 1-week.
  Interventions: Behavioral: Reminders; Behavioral: Financial Incentive
- Active Control (Active Comparator): Patients not sent any reminder message.
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Reminders — Reminders
  Arms: Message + Financial Incentive; Message Only
Behavioral: Financial Incentive — $50 financial incentive for getting vaccinated within 1-week
  Arms: Message + Financial Incentive
Other: Placebo — No special messages or incentives
  Arms: Active Control

SUMMARY:
In this work, we are assessing the impact of messaging with or without a $50 financial incentive on influenza vaccination rates in a county health system. Our main hypothesis is that a message with a $50 financial incentive will increase vaccination rates relative to a control/"treatment as usual" group. We further hypothesize that the financial incentive will increase vaccination rates relative to the message only arm.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and over
* Empaneled patients or non-empaneled patients with a primary care visit in past 18 months with valid insurance
* Due for an annual flu shot according to the electronic medical record
* Active phone number or email
* Do not have "Do not contact" flag

Exclusion Criteria:

* Under age 18
* Received an annual flu shot based on medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69972 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Vaccination status at 1 week | 1 week
  influenza vaccination status as documented in the EMR and from the California Immunization Registry (CAIRS)

SECONDARY OUTCOMES:
Vaccination status at 2 weeks | 2 weeks
  Influenza vaccination status as documented in the EMR and from the California Immunization Registry (CAIRS)
Vaccination status at 1 month | 1 month
  Influenza vaccination status as documented in the EMR and from the California Immunization Registry (CAIRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Contra Costa Health Services, Martinez, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be shared with qualified researchers upon request.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Chang TY, Jacobson M, Shah M, Pramanik R, Shah SB. Impact of reminder messages, with and without financial incentives, on influenza vaccination: A randomized trial in a California health system. Vaccine. 2026 Jan 27;75:128263. doi: 10.1016/j.vaccine.2026.128263. Online ahead of print. PMID 41604808